CLINICAL TRIAL: NCT02549612
Title: The Effect of Early Non-Surgical Treatment of Children With Middle Ear Effusion on the Hearing Level and the Health Economics
Brief Title: The Effect of Early Non-Surgical Treatment of Children With Middle Ear Effusion on the Hearing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hearing improvement after AOM
Record Dates: First submitted 2015-04-13; First posted 2015-09-15 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Secretory Otitis Media; Acute Otitis Media
Keywords: Conductive hearing loss; middle ear pressure equalization; middle ear effusion
MeSH Terms: conditions — Otitis Media with Effusion; Otitis Media; Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moniri Otovent (Experimental): A face mask is connected to a tube to which a coloured balloon is attached. The tube is also connected to ambu bag balloon. A safety valve is used to prevent too high air pressure. The ambu bag balloon is hidden in a green soft toy in the form of frog. The parent and the child hold the face mask against the mouth and the child blows the balloon. On need, mainly in the beginning of treatment course, the parent presses the frog's abdomen in order to fill the balloon with air. On the first day, a low pressure balloon is used, then it is changed with a higher pressure balloon. If no effect is noticed, (the child should experience clicking sound in one or both ears) after day 3, the balloon is replaced with a new balloon with additionally higher pressure. Full compliance for the treatment is defined as 20 blows (5 minutes) in the morning and evening for one week.
  Interventions: Device: Moniri Otovent
- Control (No Intervention): No intervention is used in this group.

INTERVENTIONS:
Device: Moniri Otovent — Please see arm description.
  Arms: Moniri Otovent

SUMMARY:
Secretory otitis media (SOM) or middle ear effusion is a common finding after acute otitis media (AOM). It is usually associated with 5-15 deci Bells hearing loss. Although spontaneous resolution with normalisation of hearing is the usual outcome, this can take several months. Secretory otitis media is the most common cause of hearing impairment in the paediatric age group. When the hearing loss caused by SOM is bilateral and persists for 3-6 months or more, surgery with tympanostomy tube insertion under general anaesthesia is indicated. In Sweden, 10000 children undergo this operation annually. Although many children with unilateral or bilateral SOM improve in the summer, the problem usually recurs in the autumn or winter. The cost of SOM for the Swedish society was 600 million Swedish crowns 2005.

In two previous studies, the investigators concluded that the nonsurgical treatment method, that was developed to assist children with SOM equalising their middle ear pressure, could normalise the hearing level in 80 % of children with SOM of minimum duration of 3 months. These children avoided therefore grommet insertion.

The investigators would like to assess the effect of this new treatment method on hearing directly after AOM. The investigators expect that using the new method could rapidly normalise hearing in these cases and thereby operation with grommet insertion could be avoided.

DETAILED DESCRIPTION:
Background:

Secretory otitis media (SOM) or middle ear effusion is the most common cause of hearing impairment in children. Hearing loss occurs due to the accumulation of fluid in the middle ear. In most of the cases, SOM follows acute otitis media (AOM). In cases when the SOM is bilateral and persists for more than 3-6 months, operation with grommet insertion under general anaesthesia is indicated. 10000 children with SOM are operated with grommet insertion every year in Sweden. In cases of unilateral hearing loss caused by SOM, grommet insertion is rarely indicated if the duration of symptoms is less than one year. Some patients develop persistent perforation in the eardrum after extrusion of the tympanostomy tube.

A new method of middle ear pressure equalisation has been developed at the Sahlgrenska University Hospital. 45 children in the age of 2-8 years with SOM that persisted for more than 3 months had been treated with this new method under the waiting period for grommet insertion. 80% of these children had been cured with regaining of normal hearing and avoided operation. No complication/side effects were noticed and the compliance was good.

Aim of the study:

To assess the effectivity of the new nonsurgical treatment method for equalisation of middle ear pressure in rapid regaining of hearing after acute otitis media in 2,5-7 years old children.

Study design:

Quantitative

Hypothesis:

Can the new nonsurgical method rapidly normalise hearing in children with middle ear effusion/secretory otitis media after acute otitis media.

Material and Method:

80 children in the age of 2,5-7 years will be offered, directly after completed treatment of AOM, inclusion in the study. All the patients will undergo during the first visit microscopic examination of the ears, audiogram and tympanogram. The children will be randomised thereafter into two groups. The first group is treated with the new method for one week. While the other group is not actively treated and will act as a control. Both groups undergo one week after randomisation new examination with microscopic examination of the ears, audiogram and tympanogram. These examinations are repeated after one and three months.

Intervention:

The first group with verified middle ear effusion after AOM is treated with the new nonsurgical method of middle ear pressure equalisation. A face mask is connected to a tube to which a coloured balloon is attached. The tube is also connected to balloon. A safety valve is used to prevent too high air pressure. A balloon is hidden in a green soft toy in the form of frog. The parent and the child hold the face mask against the mouth and the child blows the balloon. On need, mainly in the beginning of treatment course, the parent presses the frog's abdomen in order to fill the balloon with air. On the first day, a low pressure balloon is used, then it is changed to a balloon with higher pressure. If no effect is noticed, (the child should experience clicking sound in one or both ears) on the third day, the balloon is replaced with a new balloon with additionally higher pressure. Full compliance for the treatment is defined as 20 blows (5 minutes) in the morning and evening for one week.

Expected results and importance:

The investigators expect that the study will show that the new treatment method of SOM secondary to AOM can rapidly and effectively improve hearing of the affected child. This can be of great significance from medical, social and economic point of view. Hearing impairment in the paediatric age group has a great negative impact on speech development and are not only disadvantageous to the child and the parent but also for the whole society.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral middle ear effusion with resultant conductive hearing loss one week after acute otitis media.
* Intact tympanic membranes bilaterally.
* Acceptable level of written and spoken swedish language skills.

Exclusion Criteria:

* Comorbidity,
* Perforated acute otitis media or other complications of acute otitis media.

Ages: 30 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2017-03; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline (start of treatment in the treatment group or start of control in the control group) in Hearing Level measured using age suitable audiogram. | One week after baseline.
  Measuring hearing threshold using age suitable audiogram.
Change from Baseline (start of treatment in the treatment group or start of control in the control group) in Hearing Level measured using age suitable audiogram. | One month after baseline.
  Measuring hearing threshold using age suitable audiogram.
Change from Baseline (start of treatment in the treatment group or start of control in the control group) in Hearing Level measured using age suitable audiogram. | Three months after baseline.
  Measuring hearing threshold using age suitable audiogram.

SECONDARY OUTCOMES:
Change from Baseline in Middle Ear Pressure measured using tympanogram. | One week, one month and three months after baseline.
  Measuring middle ear pressure using tympanogram.
Presence of Fluid in the Middle Ear. | One week, one month and three months after baseline.
  Microscopic examination of the tympanic membrane to show the presence or absence of fluid in the middle ear.
Health Economics Measured Mainly by the Number of Parental Leave Days which the parent/parents needed to take in order to look after the child. | Three months after baseline.
Otitis Media Questionnaire-14 (OMQ-14). | Three months after baseline.
  Please see Links
Number of Health Care or Hospital Visits due to Ear Associated Problems. | Three months after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Hasse Ejnell, Study Director — Sahlgrenska University Hospital

REFERENCES:
- See also: OMQ-14 — http://www.cmaj.ca/content/suppl/2015/07/27/cmaj.141608.DC1/141608-res-3-at.pdf